CLINICAL TRIAL: NCT07058493
Title: Analgesic Effect of Using Dexmedetomidine as an Additive for (Ipack)Block in Knee Surgeries in Adult Patient; A Randomized Controlled Trial
Brief Title: Dexmedetomidine as an Additive for (Ipack)Block in Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Ismail, Associate Professor of Anesthesia, Surgical ICU and pain management at Faculty of medicine Cairo University, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: MS-491-2023
Record Dates: First submitted 2024-05-05; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Knee Surgeries
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Experimental): IPACK block with 20ml bupivacaine 0.25% alone.
  .
  Interventions: Drug: Bupivacaine
- Dexmedetomidine (Experimental): IPACK block with 20 ml of bupivacaine 0.25% with dexmedetomidine 100 μg as adjuvant.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine 100 μg as adjuvant to IPACK block with 20 ml of bupivacaine 0.25%.
  Arms: Dexmedetomidine
Drug: Bupivacaine — 20 ml of bupivacaine 0.25%.
  Arms: Bupivacaine

SUMMARY:
Dexmedetomidine used as an Additive for Ipack Block in Knee Surgery

DETAILED DESCRIPTION:
Many types of analgesia used but multimodal analgesia showed best results The interspace between the popliteal artery and capsule of the posterior knee (IPACK) block aims to blockade of sciatic nerve terminal branches for analgesia without motor affection

. (IPACK) block is a motor power sparing procedure that involves injecting local anesthetic into the space between the popliteal artery and the posterior capsule of the knee in order to treat posterior knee pain

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years
* ASA I, II .patients undergoing knee surgeries.

Exclusion Criteria:

* patient Refusal
* bleeding disorders
* skin lesion
* infection
* known allergy
* contradictions of spinal anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale at rest score during first postoperative 48 hours | 48 postoperative hours
  Visual Analog Scale at rest during first postoperative 48 hours a line 10centimeters long from zero to10 where 10 is the worst pain ever

SECONDARY OUTCOMES:
Visual Analog Scale at rest and during movement at 30 minuts, 2, 8, 16, 24, 36, and 48 hours | 48 postoperative hours
  Visual Analog Scale at rest during 48 postoperative hour a line 10centimeters long from zero to10 where 10 is the worst pain ever
Duration of the block | 48 hours
  Duration of the block
Heart Rate | 48 hours
  Heart Rate
Mean Arterial Pressure | 48 hours
  Mean Arterial Pressure
Block performance time in minutes | preoperative
  Block performance time in minutes
Incidence of adverse effects | 2 hours inPACU
  Incidence of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Dalia K Ismail, Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No